CLINICAL TRIAL: NCT00756028
Title: Short Versus Long IVF-treatment. A Prospective, Consecutive and Randomized Comparative Study
Brief Title: Short Versus Long Protocol for IVF and IVF+ICSI
Acronym: KvL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peter Hornnes, MD, DMSc (Other)
Responsible Party: Sponsor-Investigator, Peter Hornnes, MD, DMSc, MD, DMSc, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KvL
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Infertility; Ovarian Hyperstimulation Syndrome; Quality of Life; Live Birth
Keywords: OHSS; quality of life; IVF; ICSI; GnRH-agonist; GnRH-antagonist
MeSH Terms: conditions — Infertility; Ovarian Hyperstimulation Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients receiving short protocol IVF/ICSI-treatment. Intervention pharmacon: GnRH-antagonist (Orgalutran®: Ganirelix)
  Interventions: Drug: Patients receiving short protocol IVF/ICSI-treatment.
- 2 (Active Comparator): Patients receiving long protocol IVF/ICSI-treatment. Intervention pharmacon: GnRH-agonist (Synarela®: Nafarelin)
  Interventions: Drug: Long protocol

INTERVENTIONS:
Drug: Patients receiving short protocol IVF/ICSI-treatment. — Injection s.c. Orgalutran® (Ganirelix)0.25 mg once daily from day 5 of FSH-stimulation until HCG-day
  Arms: 1
Drug: Long protocol — Patients receiving long protocol IVF/ICSI-treatment. Intervention pharmacon: GnRH-agonist (Synarela®:Nafarelin)
  Arms: 2

SUMMARY:
Purpose: Comparing a GnRH agonist and an antagonist protocol for IVF/ICSI with regard to

1. frequency of ovarian hyperstimulation syndrome (OHSS) (1. outcome measure)
2. quality of life (2. outcome measure)
3. live birth rate (2. outcome measure)
4. gene expression profiles of granulosa and cumulus cells, and concentrations of estradiol and vascular endothelial growth factor in follicular fluid(not only compared between GnRH agonist and antagonist protocol, but also between patients with OHSS and no OHSS and patients becoming pregnant and not becoming pregnant (2. outcome measure), and
5. number of oocytes removed per treatment, number of embryo transfers per treatment and number of spontaneous abortions per treatment (these three parameters are tertiary outcome measures).

In addition to the above mentioned efficacy outcome measures the safety outcome measure "frequency of known side-effects" will be compared between the two protocols.

DETAILED DESCRIPTION:
Patients: 1100 patients are randomized prospectively to either treatment. Stratification: =<36 y/>36 y, IVF/ICSI, and treatment centre.

Methods: OHSS is quantified by consecutive measurements of weight, abdominal diameter, ultrasound measurements of ascites and ovarian volume, paraclinical parameters, and by a systematic patient questionnaire. Furthermore it is registered if the patients have been hospitalized and/or have had ascites drainage performed due to OHSS. Data from the first 100 patients are used together with Golans OHSS-classification, to make a more precise definition of OHSS. This definition is applied prospectively on data from the remaining patients.

Quality of life is gauged by a questionnaire. Child birth rate is ascertained by a pregnancy response questionnaire and by obtaining data from the Danish National Birth Registry.

Statistics: The study is designed to be able to show a 50% reduction of OHSS comparing short to long protocol.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for infertility receiving their first IVF or IVF+ICSI treatment

Exclusion Criteria:

* Previous IVF or IVF+ICSI-treatment
* Uterine anomalies
* It is necessary to perform direct sperm aspiration from husband's/partner's testicles
* Allergy to one of the intervention products
* Patient is 40 years or above

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1099 (Actual)
Dates: Start 2009-01; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Frequency of Ovarian Hyperstimulation Syndrome (OHSS) | 3 years

SECONDARY OUTCOMES:
Quality of life during treatment | 3 years
Live births | 3 years
Gene expression profiles of granulosa and cumulus cells | 3 years
Estradiol and vascular endothelial growth factor concentrations in follicular fluid. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Thue Bryndorf, Study Chair — Hvidovre University Hospital; Helle Meinertz, Study Chair — Hvidovre University Hospital; Peter Hornnes, Principal Investigator — Hvidovre University Hospital
Locations (2):
- Denmark (2):
  - Dronninglund Fertility Clinic, Dronninglund
  - Fertility Clinic, Hvidovre Hospital, Hvidovre

REFERENCES:
- [Derived] Toftager M, Sylvest R, Schmidt L, Bogstad J, Lossl K, Praetorius L, Zedeler A, Bryndorf T, Pinborg A. Quality of life and psychosocial and physical well-being among 1,023 women during their first assisted reproductive technology treatment: secondary outcome to a randomized controlled trial comparing gonadotropin-releasing hormone (GnRH) antagonist and GnRH agonist protocols. Fertil Steril. 2018 Jan;109(1):154-164. doi: 10.1016/j.fertnstert.2017.09.020. Epub 2017 Nov 23. PMID 29175067
- [Derived] Toftager M, Bogstad J, Lossl K, Praetorius L, Zedeler A, Bryndorf T, Nilas L, Pinborg A. Cumulative live birth rates after one ART cycle including all subsequent frozen-thaw cycles in 1050 women: secondary outcome of an RCT comparing GnRH-antagonist and GnRH-agonist protocols. Hum Reprod. 2017 Mar 1;32(3):556-567. doi: 10.1093/humrep/dew358. PMID 28130435
- [Derived] Toftager M, Bogstad J, Bryndorf T, Lossl K, Roskaer J, Holland T, Praetorius L, Zedeler A, Nilas L, Pinborg A. Risk of severe ovarian hyperstimulation syndrome in GnRH antagonist versus GnRH agonist protocol: RCT including 1050 first IVF/ICSI cycles. Hum Reprod. 2016 Jun;31(6):1253-64. doi: 10.1093/humrep/dew051. Epub 2016 Apr 8. PMID 27060174